CLINICAL TRIAL: NCT03728855
Title: A Multicentre Study on the Effects of Self-administration of Medication During Hospitalization on Medication Safety, Adherence, and Patient Satisfaction in Dutch Hospitals
Brief Title: Effects of Self-administration of Medication During Hospitalization on Medication Safety, Adherence, and Patient Satisfaction in Dutch Hospitals
Acronym: MIEB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult recruitment, despite several interventions.
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: UMCN-AKF-18.02
Record Dates: First submitted 2018-10-05; First posted 2018-11-02 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Medication Safety; Patient Safety; Patient Empowerment
Keywords: Self-administration of medication; SAM; Medication Safety; Patient Empowerment; Patient Satisfaction; Staff Satisfaction
MeSH Terms: conditions — Patient Participation; Patient Satisfaction | interventions — Self Administration

STUDY DESIGN:
Intervention Model Description: The intervention of this study is the implementation of self-administration of medication (SAM) by hospitalized patients. SAM will be compared to standard care.
Who Masked: Outcomes Assessor
Masking Description: The subject, staff and investigators are aware of which method of medication administration the patient is given, SAM or standard care. Only the data analysis is blinded by anonymizing and coding all data. Furthermore, an independent person will perform the data analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Based on an (electronic) order placed by a physician, nurses collect medication and provide patients with the ordered medication in a timely matter. Nurses document the administration either in an electronic medical record or on paper.
- Self-administration of medication (SAM) (Experimental): During SAM medication is stocked at the patient's bedside. When medication is scheduled to be administered, patients collect those form their own stock, administer, and document the administration by themselves. Once daily nurses check whether patients succeeded in administration for all prescriptions of the last 24 hours. Each day, patients are qualified for SAM. In the case patients do not meet the criteria of SAM, they will be excluded from SAM.
  Interventions: Behavioral: Self-administration of medication (SAM)

INTERVENTIONS:
Behavioral: Self-administration of medication (SAM) — Patients use medication from their own stock, self-administered.
  Arms: Self-administration of medication (SAM)

SUMMARY:
During hospitalization, medication administration errors (MAEs) occur daily in health care and can lead to serious harm. Improvement of medication safety is a major concern to policymakers and health care workers. Inpatient self-administration of medication (SAM) during hospital admission could be a way to reduce MAEs. Therefore the aim of this study is to determine the effect of inpatient self-administration of medication on the number of medication administration errors during hospitalization.

DETAILED DESCRIPTION:
Objective: the main objective of this study is to determine the effect of inpatient self-administration of medication on the number of medication administration errors during hospitalization. The secondary objectives of this study are to determine:

1. The effect of inpatient self-administration of medication on the severity of medication administration errors during hospitalization
2. The effect of inpatient self-administration on medication adherence after hospitalization
3. The effect of inpatient self-administration of medication on patient satisfaction during hospitalization
4. The effect of inpatient self-administration of medication on staff satisfaction during hospitalization

Study design: multicentre prospective quasi-experimental study with a pre-post design

Study population: hospitalized ≥ 16 years old patients

Intervention: the implementation of self-administration of medication by hospitalized patients. SAM will be compared to standard care.

Main study parameters: The primary outcome measure of the study is the proportion of medication administrations with one or more medication administration errors (MAEs). Secondary outcome measures will be: severity of MAEs, medication adherence after hospitalization, patient satisfaction during hospitalization, and staff satisfaction. For all outcome measures the effect of SAM will be compared to standard care.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: all subjects have to fulfil two questionnaires, one during hospitalization and one approximately three months after leaving the studied ward, e.g. hospital discharge or transfer. The subjects that are included in de post study period have to self-administrate medication that's suitable for SAM. The risk of SAM during hospitalization is estimated as the risk patients are at home when using medication. The burden of SAM is classified as low because results of a recent questionnaire shows that admitted patients have the urge to act in SAM schemes.

ELIGIBILITY:
Inclusion Criteria:

* All patients (≥ 16 years old) admitted to the ward who use medication or will be using medication at home after hospital discharge and are able to administer (part of) this medication themselves

Exclusion Criteria:

* Not providing informed consent
* The use of a medication box without original medication boxes
* The use of medication pre-packaged by automated dispensing system
* The need of homecare support to administer medication
* The need of an informal caretaker to help with medication administration
* Admitted from a nursing home and medication is under supervision of the staff
* Not understanding the Dutch language, written or spoken
* The subject is not capable of managing SAM (due to mental or physical state)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Proportion of medication administration errors | 2 weeks
  The doctor's prescriptions as noted in the CPOE system will be compared to the observed medication administration and any discrepancy will be marked as an MAE. The number of erroneous medication administrations (containing 1 or more errors) will be divided by the number of observed drug administrations plus the number of omissions (concept of opportunities).

SECONDARY OUTCOMES:
Severity of MAEs | 2 weeks
  Severity of MAEs will be determined by two healthcare professionals, a physician and a pharmacist.To classify the severity of MAEs the NCC MERP Index for categorizing medication errors will be used. Thereafter consensus will be reached. The experts will be blinded to the period (usual care or intervention) during which the problem occurred.
Medication adherence after hospitalization | 3 months
  Medication adherence after hospitalisation will be measured using the Medication Adherence Reasons Scale (MAR-Scale). The MAR-Scale measures medication non-adherence based on the reasons for non-adherence so that each reason can be matched with a corresponding intervention. Approximately three months after hospitalization, a questionnaire consisting of six questions concerning the patient's medication use will be sent to all included patients by email.
Medication adherence after hospitalization | 1 year
  With the use of the pharmacy refill dates the Medication Refill Adherence (MRA) is calculated.
  - 1 year after inclusion: pharmacy refill data will be collected
Patient satisfaction during hospitalization | 7 days
  Patient satisfaction will be measured by the visual analogue scale (VAS) for patient satisfaction.
Patient satisfaction during hospitalization | 7 days
  Patient satisfaction will be measured by the Beliefs about Medicine Questionnaire (BMQ).
Staff satisfaction | 1 year
  Staff satisfaction will be measured using The Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM). These are four-item measures of implementation outcomes that are often considered "leading indicators" of implementation success. These measures can be administered to a wide range of stakeholders to determine the extent to which they believe an intervention or an implementation strategy is acceptable, appropriate, and feasible. At the end of the study hospital staff will be asked to complete the questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Bart van den Bemt, PharmD, PhD, Principal Investigator — Radboudumc/ Sint Maartenskliniek
Locations (8):
- Netherlands (8):
  - Radboudumc, Nijmegen, Gelderland
  - Sint Maartenskliniek, Ubbergen, Gelderland
  - MUMC+, Maastricht, Limburg
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - ETZ, Tilburg, North Brabant
  - Groene Hart Ziekenhuis, Gouda, South Holland
  - Meander Medisch Centrum, Amersfoort